CLINICAL TRIAL: NCT00629551
Title: An Eight-week, Double-blind Study to Evaluate the Efficacy, Safety, and Tolerability of Two Fixed Doses of Saredutant (100 mg and 30 mg) Once Daily in Combination With Paroxetine 20 mg Once Daily Compared to Saredutant Placebo in Combination With Paroxetine 20 mg Once Daily in Patients With Major Depressive Disorder
Brief Title: An Eight-week Study of Saredutant and Paroxetine as Combination Treatment for Major Depressive Disorder
Acronym: COMPASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10438; EudraCT 2007-003863-31
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; Depression; Major Depressive Episode; Antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — SR 48968; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Saredutant 100mg and Paroxetine 20 mg (Experimental): combined saredutant 100mg and paroxetine 20mg once daily for a maximum of 8 weeks
  Interventions: Drug: saredutant (SR48968); Drug: paroxetine
- Saredutant 30mg and Paroxetine 20mg (Experimental): combined saredutant 30mg and paroxetine 20mg once daily for a maximum of 8 weeks
  Interventions: Drug: saredutant (SR48968); Drug: paroxetine
- Paroxetine 20 mg and saredutant placebo (Active Comparator): paroxetine 20mg and saredutant placebo once daily for a maximum of 8 weeks
  Interventions: Drug: paroxetine; Drug: placebo
- Placebo (Placebo Comparator): Saredutant placebo and paroxetine placebo once daily for one week during screening period and maximum of 8 weeks for the active phase
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: saredutant (SR48968) — oral administration,capsules
  Arms: Saredutant 100mg and Paroxetine 20 mg; Saredutant 30mg and Paroxetine 20mg
Drug: paroxetine — oral administration, capsules
  Arms: Paroxetine 20 mg and saredutant placebo; Saredutant 100mg and Paroxetine 20 mg; Saredutant 30mg and Paroxetine 20mg
Drug: placebo — oral administration, capsules
  Arms: Paroxetine 20 mg and saredutant placebo; Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of saredutant 100mg or 30mg once daily in combination with paroxetine 20mg once daily compared to saredutant placebo in combination with paroxetine 20mg once daily in patients with major depressive disorder. The study also includes a double-placebo group (saredutant placebo in combination with paroxetine placebo).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with recurrent Major Depressive Disorder

Exclusion Criteria:

* Symptoms of current depressive episode for less than 30 days or more than 2 years
* Mild depression, as measured by standard clinical research scales
* Significant suicide risk
* Lack of sexual activity (including masturbation)
* Other psychiatric conditions that would obscure the results of the study
* History of failure to respond to antidepressant treatment
* Pregnancy or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Hamilton Depression Rating Scale (HAM-D) total score | 8 weeks
Change from Baseline in the Changes in Sexual Functioning Questionnaire (CSFQ) total score | weeks

SECONDARY OUTCOMES:
Change from baseline in the Clinical Global Impression severity of illness score | 8 weeks
Change from baseline in the HAM-D depressed mood item scores | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (8):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea